CLINICAL TRIAL: NCT07176949
Title: Project on Myopia Surveillance and Intervention Services for Preschool Children in Shanghai
Brief Title: Early-Onset Myopia Intervention Project
Acronym: EOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-20240712-11
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Pre-myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention (No Intervention): No intervention for myopia control
- Spectacle Lenses with Highly Aspherical Lenslets (Experimental): Wearing spectacle lenses with highly aspherical lenslets for myopia control
  Interventions: Device: Spectacle lenses with highly aspherical lenslets
- 0.01% Atropine (Experimental): Nightly use of 0.01% atropine eyedrops for myopia control
  Interventions: Drug: 0.01% atropine eye drops
- 0.05% Atropine (Experimental): Nightly use of 0.05% atropine eyedrops for myopia control
  Interventions: Drug: 0.05% atropine eye drops

INTERVENTIONS:
Drug: 0.01% atropine eye drops — Participants will use 0.01% atropine eyedrops nightly for myopia control.
  Arms: 0.01% Atropine
Drug: 0.05% atropine eye drops — Participants will use 0.05% atropine eyedrops nightly for myopia control.
  Arms: 0.05% Atropine
Device: Spectacle lenses with highly aspherical lenslets — These are a special type of eyeglass lenses designed primarily to slow down the progression of myopia (nearsightedness) in children. The center of the lens provides a clear correction for distance vision, just like regular glasses. The surrounding area contains hundreds of tiny, invisible, and highly aspherical (complex curved) microlenses. These microlenses create a special optical effect. While the child looks straight ahead clearly, peripheral light rays are focused in front of the retina. This is called "myopic defocus." Research suggests that this myopic defocus signal helps to control the excessive elongation of the eyeball, which is the main cause of myopia getting worse.
  Arms: Spectacle Lenses with Highly Aspherical Lenslets

SUMMARY:
The prevalence of myopia among children has been increasing year by year, which has become a globle public health issue. Studies have shown that defocusing lenses and atroping eyedrops can control the progression of myopia, but there is little evidence of its efficacy in myopia intervention of young pre-schoolers who will face a greater risk of progression to high myopia later in life. Therefore, this study aims to evaluate the effectiveness and safety of spectacle lenses with highly aspherical lenslets (Essilor's Stellest) , as well as 0.01% and 0.05% low concentration atropine eyedrops in myopia intervention among young children aged 3-6.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-6 years, gender unrestricted;
* Bilateral cycloplegic spherical equivalent (SE) ≤ +0.75 D, astigmatism ≤-2.5 D, anisometropia ≤2.5 D;
* Best corrected visual acuity: ≥0.5 for ages 3-5, ≥0.7 for age 6;
* Accept regular follow-up, written informed consent from guardians, verbal informed consent from children;
* Possess normal thinking and language communication skills, and can actively cooperate to wear spectacles as required.

Exclusion Criteria:

* Existence of strabismus or amblyopia or other binocular vision abnormalities, accommodation dysfunction, cataract and history of eye surgery;
* Any ocular or systemic disease that may affect vision and refractive development (e.g., Keratoconus, Marfan syndrome, retinopathy of prematurity, etc.);
* Current or previous use of other treatments for myopia intervention, such as pharmacological (atropine) and optical (orthokeratology lenses or DIMS spectacle lenses) approaches, interrupt use for at least 4 weeks;
* Allergy or contraindication to cycloplegic drugs;
* Epilepsy or other mental disorders unable to expressing consent;
* Other conditions deemed unsuitable for participation by the researcher.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 508 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cycloplegic spherical equivalence | 2 year
  Measured by an auto-refractometer

SECONDARY OUTCOMES:
Changes in axial length | 2 years
  Measured by an IOL-Master
Proportion of subjects with non-rapid myopia progression | 2 years
  Rapid myopia progression is defined as: spherical equivalence increase (become less positive or more negative refractive error) of any eye ≥ 0.5 D in half a year.
The duration of non-rapid myopia progression | 2 years
  Rapid myopia progression is defined as: spherical equivalence increase (become less positive or more negative refractive error) of any eye ≥ 0.5 D in half a year.

OTHER OUTCOMES:
Changes in choroid/retina thickness | 2 years
  Measured by SS-OCT
Changes in BCVA | 2 years
  Best corrected visual acuity
Changes in IOP | 2 years
  Intraocular pressure
Changes in AMP | 2 years
  Amplitude of Accommodation
Changes in Stereopsis | 2 years
  Using Titmus Fly Test
Changes in TBUT | 2 years
  Tear Film Break-Up Time
Changes in anterior segment parameters | 2 years
  Measured by Pentacam
Changes in Hemodynamic Parameters of the Ocular Fundus | 2 years
  Measured by SS-OCTA
Compliance indicators | 2 years
  Daily wearing duration, wearing habits and patterns, frequency of eye drops use.
Side Effects and Adverse Events | 2 years
  Incidence of glare, diplopia, blurred vision, photophobia, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, Shanghai Municipality, China